CLINICAL TRIAL: NCT06649994
Title: Transcranial Magnetic Stimulation and Inhibitory Control Training to Reduce Binge Eating: Brain and Behavioral Changes (BE-NEMOIC)
Brief Title: Transcranial Magnetic Stimulation and Inhibitory Control Training to Reduce Binge Eating: Brain and Behavioral Changes
Acronym: BE-NEMOIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Raquel Vilar López (Other)
Collaborators: Junta de Andalucia (Other Government)
Responsible Party: Sponsor-Investigator, Raquel Vilar López, Principal Investigator, Universidad de Granada
Organization: Universidad de Granada (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ProyExcel_00776
Record Dates: First submitted 2024-09-17; First posted 2024-10-21 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Binge Eating; Inhibition, Psychological
Keywords: binge eating; rTMS; inhibitory control; training
MeSH Terms: conditions — Bulimia; Inhibition, Psychological

STUDY DESIGN:
Intervention Model Description: Parallel group randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The psychologists that conduct the assessments (screening, assessment sessions and follow-ups) will be blinded to the group allocation during the whole project. Further, all participants will be blind to their condition. Also, the people who perform the statistical analyses will be blind to the condition of the groups, through the coding of the interventions. Only the therapist performing the interventions will not be blind to the allocation of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active iTBS of the DLPFC (Experimental): The experimental group will: i) receive an informative session; ii) 2 sessions of pre-treatment assessment (one with fMRI and one with questionnaires); iii) participate in 10 daily individual intervention sessions that consist of iTBS of the left dlPFC followed immediately inhibitory control training, that will last about 10-20 minutes each; iv) 2 sessions of post-treatment assessment (one with fMRI and one with questionnaires); v) one follow-up assessment session three months after completing the intervention
  Interventions: Device: Active iTBS of the DLPFC; Behavioral: Computerized inhibitory control training
- Active iTBS of the vmPFC (Experimental): The experimental group will: i) receive an informative session; ii) 2 sessions of pre-treatment assessment (one with fMRI and one with questionnaires); iii) participate in 10 daily individual intervention sessions that consist of iTBS of the vmPFC followed immediately by inhibitory control training, that will last about 10-20 minutes each; iv) 2 sessions of post-treatment assessment (one with fMRI and one with questionnaires); v) one follow-up assessment session three months after completing the intervention
  Interventions: Device: Active iTBS of the vmPFC; Behavioral: Computerized inhibitory control training
- Active Control (Placebo Comparator): The active control group will: i) receive an informative session; ii) 2 sessions of pre-treatment assessment (one with fMRI and one with questionnaires); iii) participate in 10 daily individual intervention sessions that consist of iTBS of the vertex (sham) followed immediately by inhibitory control training, that will last about 10-20 minutes each; iv) 2 sessions of post-treatment assessment (one with fMRI and one with questionnaires); v) one follow-up assessment session three months after completing the intervention
  Interventions: Device: iTBS of the vertex (sham); Behavioral: Computerized inhibitory control training

INTERVENTIONS:
Device: Active iTBS of the DLPFC — Participants will receive a 3 minutes intermittent Theta Burst Stimulation of the DLPCF of the left hemisphere while not performing any other task
  Arms: Active iTBS of the DLPFC
Device: Active iTBS of the vmPFC — Participants will receive a 3 minutes active intermittent Theta Burst Stimulation of the vmPFC while not performing any other task
  Arms: Active iTBS of the vmPFC
Device: iTBS of the vertex (sham) — Participants will receive a 3 minutes active intermittent Theta Burst Stimulation of the vertex while not performing any other task
  Arms: Active Control
Behavioral: Computerized inhibitory control training — Participants will perform the task of the FoodT app for 10 minutes immediately after iTBS (taking advantage of time of maximum brain potentiation, Rossi et al., 2009).
  This task pairs high-calorie meals with the no-go cue. Images appear on the left, right or center of the smartphone screen and they must touch it or not (depending on the cue) with their index finger as quickly as possible. Participants earn points for correct tap responses and lose points for incorrect tap responses: If the image has a green border around it, you must tap the image and win 1 point. But if the image has a red border around it, you must inhibit the tapping response or you will lose 1 point. Participants must respond as quickly and accurately as possible and improve reaction time.
  Pictures of healthy and unhealthy foods are always paired with the Go and the No-Go signal, respectively. Non-food images are paired 50% of the time with the Go and the No-Go signal
  Other Names: FoodT

SUMMARY:
People with BE are characterized by high impulsivity, high levels of craving for high-calorie foods, deficits in inhibitory control, and maladaptive decision making. These characteristics are related, at brain level, to alterations in the activation of areas such as the dorsolateral prefrontal cortex (DLPFC) and ventromedial prefrontal cortex (vmPFC) among other brain areas and their connectivity. The investigators propose an intervention that seeks to target these issues. Thus, the present study aims to characterize the effects of neuromodulation with intermittent theta burst stimulation (iTBS) of the DLPFC or the vmPFC in combination with inhibitory control training to produce brain, cognitive and behavioral changes, and modify altered biological parameters in people with BE. Participants will be randomly allocated to one of three groups: 1) a group that will receive active iTBS of the DLPFC together with inhibitory control training with a food Go/NoGo paradigm, and 2) a group that will receive active iTBS of the vmPFC together with inhibitory control training with a food Go/NoGo paradigm, and 3) an active control group that will receive sham iTBS together with inhibitory control training with a food Go/NoGo paradigm. The investigators hypothesized that neuromodulation with iTBS applied to DLPFC or vmPFC will modify the dynamics of different brain circuits associated with binge eating. Neuromodulation of the DLPFC or vmPFC in combination with inhibitory control training, will be associated with: (i) decreased appraisal of unhealthy foods, (ii) reduced food craving, (iii) improved eating behavior, (iv) modified brain connectivity and activation both at rest and linked to task performance with food stimuli, (v) a decrease in the frequency and intensity of binge eating, (vi) improved emotional symptoms and emotional eating (depression, anxiety, emotional regulation, emotional eating, reward-related eating, non-homeostatic eating), (vii) improved cognitive abilities (motor and cognitive inhibition, delay of gratification, impulsivity, working memory, cognitive flexibility and decision making), (viii) changes in biological parameters associated to the interventions (plasma and microbiota), and (ix) advantages in cost-effectiveness and cost-utility based on economic evaluation analyses.

DETAILED DESCRIPTION:
1. STARTING HYPOTHESES AND GENERAL OBJECTIVE HYPOTHESIS: Neuromodulation with intermittent theta burst stimulation (iTBS) applied to the left dorsolateral prefrontal cortex (DLPFC) or the ventromedial prefrontal cortex (vmPFC) in combination with inhibitory control training with a food Go/NoGo paradigm, will be associated with: (i) decreased appraisal of unhealthy foods, (ii) reduced food craving, (iii) improved eating behavior, (iv) modified brain connectivity and activation both at rest and linked to task performance with food stimuli, (v) a decrease in the frequency and intensity of binge eating, (vi) improved emotional symptoms and emotional eating (depression, anxiety, emotional regulation, emotional eating, reward-related eating, non-homeostatic eating), (vii) improved cognitive abilities (motor and cognitive inhibition, delay of gratification, impulsivity, working memory, cognitive flexibility and decision making), (viii) changes in biological parameters associated to the interventions (blood and microbiota), and (ix) advantages in cost-effectiveness and cost-utility based on economic evaluation analyses.

GENERAL OBJECTIVE: To determine the effects of neuromodulation with iTBS in DLPFC or vmPFC in combination with inhibitory control training to generate brain, behavioural, emotional, cognitive and biological changes in people with binge eating (BE).

1.1. Specific Aims: Objective 1: To study the differential effect of iTBS applied to the left DLPFC compared to vmPFC and sham iTBS (applied to vertex), in combination with inhibitory control training, for the treatment of people with binge eating (improvements in frequency and intensity of binge eating, craving, eating behavior, emotional symptoms and emotional eating, cognitive measures and biological parameters).

Objective 2: To characterize the effects of neuromodulation with iTBS of DLPFC or vmPFC, in combination with inhibitory control training to modify brain connectivity and activation both at rest and linked to task performance with food stimuli with functional magnetic resonance imaging (fMRI).

Objective 3: To determine the relationship of biological parameters obtained in blood, saliva, urine and faeces, as well as candidate genes, with neuropsychological variables (depression, anxiety, stress, emotional regulation, emotional eating, craving, motor and cognitive inhibition, food valuation, delay of gratification, impulsivity, working memory, flexibility and decision making) and brain neuroimaging (activation, grey and white matter volume, connectivity).

Objective 4: To analyze the economic evaluation of the cost-effectiveness and cost-utility of combined training (neuromodulation with iTBS and inhibitory control training) in people with BE, and to analyze the budgetary impact of the program if it was implemented in the public health system.

METHODOLOGY

2.1. Design: Randomized controlled trial of parallel groups.

2.2. Participants: Participants (N=150) will be randomly allocated to three groups: (i) group 1 (active stimulation of the DLPFC with iTBS and inhibitory control training) n=50; (ii) group 2 (active stimulation of the vmPFC with iTBS and inhibitory control training) n=50; group 3 (active control group of sham iTBS and inhibitory control training) n=50.

2.3. Interventions: Pre-treatment interventions (all groups). First, all participants will participate in a group briefing informational session about the study. Also, informative videos and brochures will be provided. In this session no nutritional and exercise recommendations will be given.

Intervention (experimental and active control groups). Duration: 2 weeks of 5 daily sessions of about 10-20 minutes. Sessions have two parts:

Part 1. Neuromodulation with iTBS (DLPFC or vmPFC or vertex) (3 minutes net time) Part 2. Inhibition training with the Food Trainer task (10 minutes net time)

2.4. Outcome measures: binge eating symptoms and food craving-stait will be the main outcome measures. Secondary outcomes will measure changes in neuroimaging measures (brain connectivity at rest, food go/no-go paradigm and food decision making tasks), changes in eating behavior, changes in emotional symptoms and emotional eating (depression, anxiety, stress, emotion regulation, emotional eating, reward-related eating, non homeostatic eating), biomarkers and cognitive measures. Exploratory variables will include sociodemographic information, previous treatments, motivation for change, and biological and clinical variables. Further, assessment will include screening and descriptive variables, and measures to calculate cost-effectiveness, cost-utility and budget impact of the intervention program.

1. PROCEDURE Assessments will be delivered online through LimeSurvey and Milliseconds platforms. Inclusion and exclusion criteria will be checked through the data collected in a questionnaire of sociodemographic and clinical variables. Further, psychopathology exclusion criteria will be tested with three questionnaires to measure depression, anxiety, and stress symptoms as well as severity of binge eating episodes (BDI, DASS-21 and QEWP-5), and a short clinical interview by phone and/or information requested by email in those cases where there are doubts about any of the aspects collected through the online instruments.

All candidates who meet the criteria will attend an information meeting about the project in which participants will receive written and oral information and will be asked for their informed consent. Then, participants will be randomly assigned to groups before the pre-treatment assessment sessions. A simple randomization will be performed by generating five-letter codes with Calculado.net and randomizing the codes into three different groups using Rafflys. The three groups of the study will complete all the three assessments (pr, post and 3-month follow-up). What will differentiate the groups will be, therefore, the stimulation area: active iTBS applied to the left DLPFC with inhibitory control training vs. active iTBS applied to the vmPFC with inhibitory control training vs. sham iTBS (applied to the vertex) with inhibitory control training. At the end of the project, if one treatment is more effective, the other two groups will be offered the complete treatment sessions.

Informative and assessment sessions will be developed in groups of 4-6 people through the platform GoogleMeet. iTBS sessions will be administered individually. If a participant misses a session, it will be rescheduled for the beginning of the next week at a similar time. There will be at least 10 experimental groups of DLPFC stimulation intervention combined with inhibitory control training (50 participants), 10 experimental groups of vmPFC stimulation intervention combined with inhibitory control training (50 participants), and 10 active control groups of sham stimulation (50 participants). The program will comprise 5 weeks including two assessments (pre- and post-treatment), ten intervention sessions (two weeks of 5 daily sessions), and one information session. Also, a follow-up will be conducted 3 months after treatment (see below). Assessment sessions will last about 2 hours while intervention sessions will be approximately 10 to 20 minutes. Sessions will consist of the following:

1. Informative session (session 1; week 1): For the participants to understand the foundation of the intervention, participantes will be informed about the aims, basis of the project and the procedure of the research. Participants will be provided written informed consent as well. At the end of this session, participants will be asked for their informed written consent.
2. Pre-treatment assessment (session 2 and 3; week 2): All participants will complete, in session 1, the following instruments to assess the main and secondary outcomes, and the exploratory and economic measures: WCST, Food Go/NoGo, IGT, Stroop, Food DD, N-Back, CFA, DASS-21, BDI-II, PEMS, RED, DEBQ, PSRSQ, ERQ, UPPS-P, SF-36, SOCRATES 00, QEWP-5, sociodemographic questionnaire and questions about used health resources. Also, all participants will undergo the fMRI session (session 2) and biological sample collection (blood, saliva, feces and urine)
3. Intervention sessions (sessions 4 to 13; weeks 3 and 4): Intervention will consist of five weekly individual sessions for two weeks, with a 10-20 minutes total duration each. The stimulation parameters are based on the protocols for the application of iTBS in people with food intake problems, and following international safety recommendations.

   The procedure in the three groups consists of:

   i) Localization of the stimulation area by T1 sequence structural neuroimaging images using the Brainsight software for the correct placement of the stimulation coil: in the active stimulation groups it will be the left DLPFC area (x -37, y -34, z 78) corresponding to F3 position on the 10-20 EEG system or the vmPFC area (x -24, y 66, z 12) corresponding to FP1 position on the 10-20 EEG system. In the control group it will be the vertex (x 0, y-34, z 78), an area without cognitive effects after stimulation but matching the sensory effects. After that, neuromodulation with iTBS for 3 minutes with parameters of: frequency 50 Hz, number of pulses 3; number of bursts 10; cycle duration 8 seconds; number of cycles 20; burst frequency 5 Hz; and total number of pulses 600. The stimulation intensity will be maintained at 30% of the stimulator's maximum output.

   ii) Cognitive inhibitory control training (10 minutes): It will be performed with the Food T app, for 10 minutes and will be applied immediately after the iTBS, taking advantage of its time of maximum brain potentiation. In this application, the task consists of touching as quickly as possible the items that appear surrounded with a green circle, and not responding to the items surrounded by a red circle. Some images correspond to food and others are not related to food. Participants can select the categories of the images participants want to train, which should correspond to the foods used for binge eating (candy/gummies, cakes, chocolate, cookies, alcohol, chips, bread, cheese, fast food - burgers, take-out food -, sweet sodas, meat, pizza). Inhibitory control training consists of pairing high-calorie foods 100% of the time with the No-Go signal.
4. Post-treatment assessment (session 14 and 15, week 5): To evaluate the effectiveness of the interventions, BMI and craving (FCQ-T/S-r) will be registered (main outcomes), and the following instruments will be administered to obtain the secondary outcomes; WCST, Food Go/NoGo, IGT, Stroop, Food DD, N-Back, CFA, DASS-21, BDI-II, PEMS, RED, DEBQ, PSRSQ, ERQ, UPPS-P, SF-36 and questions about used health resources. Also, fMRI and biological samples of the pre-treatment assessment will be repeated.
5. Follow-up (sessions 16; week 15): Follow-up at 3 months after the intervention will include the following measures: WCST, Food Go/NoGo, IGT, Stroop, Food DD, N-Back, CFA, DASS-21, BDI-II, PEMS, RED, DEBQ, PSRSQ, ERQ, UPPS-P, SF-36, and interview about used health resources sociodemographic questionnaire and questions about used health resources and collection of biological samples and anthropometric measures to obtain the main and secondary outcome measures. Every month after the end of the treatment, participants will be contacted by email and mobile message to maintain adherence.

Participants will be instructed to eat two hours before all evaluations (pre- and post-treatment, and the follow-up) and iTBS sessions. All the assessments will be carried out at the same hour.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 20 and 39.9
* Age between 18 and 60 years
* Two or more binge eating episodes in the past month (assessed with the Binge Eating Scale)
* Proficiency in the Spanish language
* Right lateral dominance to avoid differential effects due to cortical hemispheric specialization

Exclusion Criteria:

* Traumatic, digestive, metabolic or systemic disorders that affect the central nervous system, autonomic or endocrine
* Psychopathological disorders or presence of severe symptoms in the Depression Anxiety and Stress Scale-21 (DASS-21)
* Eeating disorders other than Binge Eating Disorder, or severe or extreme Binge Eating Disorder (8 or more binges per week)
* Contraindication for performing functional magnetic resonance imaging (pregnancy, metal implants, etc.) or iTBS (tinnitus, dizziness, surgical interventions, diseases or drugs that affect the central nervous system, etc.).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Binge eating symptoms | Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17)
  The Binge Eating Scale (BES) is a self-administered questionnaire composed of 16 items: eight items that describe behavioral manifestations (for example, eating fast or consuming large amounts of food) and eight items on associated feelings and cognitions (for example, fear of not stopping eating). Each item has a response range from 0 to 3 points (0 = no severity of the symptom, 3 = serious problems on the symptom)
Food craving | This will be measured in Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17)
  The Food Craving Questionnaire Stait-reduced (FCQ-S-r) will be administered to obtain the total score, indicative of the craving state at the time of the evaluation.

SECONDARY OUTCOMES:
Changes in Food decision making (neuroimaging measures) | From baseline (week 2) to the end of the treatment (week 5)
  The task that will be used, consists of three phases: two rating phases and one decision phase with 50 food images. Participants have to answer on a 5-point Likert scale how healthy they consider the food to be (block 1) and how much they like the taste of the food (block 2). In the third block, the participant decides whether they prefer to eat a neutral reference food (calculated from the previous two blocks) or an alternative food. These forced choices lead to cognitive conflict when the reference food is considered tastier and the alternative food healthier or vice versa. Among trials with cognitive conflict, the choice of the healthier food is defined as a controlled choice, and the choice of the tastier food as an uncontrolled choice. Activation will be compared between the controlled vs. uncontrolled choice conditions.
  The task will be analysed to assess the brain activity associated with the task, using a psychophysiological interaction analyses (PPI).
Changes in Brain connectivity at rest (neuroimaging measures) | From baseline (week 2) to the end of the treatment (week 5)
  Participants will be instructed to remain still, with their eyes closed, trying not to think about anything in particular for 9 minutes to obtain images to study the resting connectivity of different brain networks. On the one hand, an independent component analyses (ICA) will be performed, which will allow comparison of the different brain networks, as a whole, between the groups, with special interest in those that have been shown to be altered in the PD population. On the other hand, seed-based connectivity analyses will be performed, in which changes in functional connectivity between the CPFDL and the rest of the brain will be observed.
Changes in White matter integrity (neuroimaging measures) | From baseline (week 2) to the end of the treatment (week 5)
  Participants will be asked to remain still for 10 minutes to obtain diffusion tensor imaging (DTI) which provides indirect measurements of the architecture and connectivity of white matter fibres. The study of the DTI images will be carried out with the FSL programme, which allows the integrity of the white matter of the different groups to be measured by evaluating the fractional anisotropy (FA) and apparent diffusion coefficient (ADC) maps.
Changes in Food Go/No-go Paradigm (neuroimaging measures) | From baseline (week 2) to the end of the treatment (week 5)
  Activation during Go and No-go items will be calculated according to the type of images (high calorie and low-calorie foods).
Changes in eating behavior | From baseline (week 2) to the end of the treatment (week 5) and follow-up (week 17)
  Eating behavior: Diet information during the last year (pre-treatment), two last weeks (post-treatment) and tree last months (follow-up) will be collected through a validated food frequency questionnaire (CFA) with 52 items in which participants must record quantities of all the foods and drinks they had consumed during those periods. These data will be transformed into the number of total calories ingested, as well as the number of calories from fats, carbohydrates, and sugars.
Anxiety and Stress. Mean change from baseline at post-intervention | From baseline (week 2) to the end of the treatment (week 5) and follow-up (week 17)
  The Depression Anxiety Stress Scale-21 (DASS-21) will be used, taking into account scores on the stress and anxiety subscales. The scores for both subscales range from 0 to 21, a higher score indicating higher anxiety or stress
Depression symptoms. Mean change from baseline at post-intervention | From baseline (week 2) to the end of the treatment (week 5) and follow-up (week 17)
  Depression symptoms will be measured with the BDI-II.This scale is asses severity of depression. The scores range from 0 to 63 points. The higher the score, the greater the severity of depressive symptoms
Non homeostatic eating. Mean change from baseline at post-intervention | From baseline (week 2) to the end of the treatment (week 5) and follow-up (week 17)
  Dutch Eating Behaviour Questionnaire (DEBQ): it will be administered to assess restrictive eating behaviours related to external cues and emotional states. Higher scores in each subscale reflect higher level of restrained, emotional, and external eating, respectively.The DEBQ uses a 5-point Likert scale, ranging from never (1) to very often (5). The average score is calculated for each subscale by adding scores obtained from individual items and dividing them by the number of items included in a subscale (mean range: 1-5).
Reward-related eating. Mean change from baseline at post-intervention | From baseline (week 2) to the end of the treatment (week 5) and follow-up (week 17)
  Reward-related eating. Reward-Based Eating Scale (RED): it is a 13 items questionnaire that assess worries about foods, losing intake control and absence of satiety. Higher scores reflect higher reward-based eating drive.
Emotional eating. Mean change from baseline at post-intervention | From baseline (week 2) to the end of the treatment (week 5) and follow-up (week 17)
  Emotional eating. Coping subscale of the Palatable Eating Motives Scale (PEMS): it will be used to evaluate the intentionality for eating palatable foods to face negative emotions. The coping subscale includes items that are scored on a 5-point Likert-type scale, the total range being from 5 to 25 points. Low scores indicate that the person rarely resorts to the consumption of pleasant foods as a strategy to cope with negative emotions or stressful situations. High scores suggest that the person frequently uses palatable food as a strategy to cope with stress or negative emotions, which may be related to unhealthy eating habits or emotional eating patterns.
Emotion Regulation Strategies. Mean change from baseline at post-intervention | From baseline (week 2) to the end of the treatment (week 5) and follow-up (week 17)
  Emotion Questionnaire (ERQ): It examines emotional regulation strategies. It10 items to examine cognitive reappraisal and expressive suppression strategies. In cognitive reappraisal the highest score (42) is associated with better emotional outcomes while in expressive suppression the highest score (28) is linked to poorer well-being. Each item is rated on a Likert scale from strongly disagree (1) to strongly agree (7).
Motor inhibition. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17)
  Motor inhibition: FoodT app will register reaction time and commission errors. In the FoodT app reaction time for the high-calorie and low-calorie foods paired with the go and the no-go signal. The average response time for go and no-go items will be calculated according to the type of images (appetizing and healthy foods), and commission errors will be recorded.
Cognitive inhibition. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17)
  Cognitive inhibition: Food Stroop Task. Using a Stroop task with food, the interference of food-related words on task performance can be measured as an assessment of cognitive inhibition.
Delay of gratification. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17)
  Delay of gratification: Food Delay Discounting (Food DD). Score on the Food Delay Discounting will be used to measure the sensitivity to immediate rewards vs higher value rewards delayed. Participants' choices are recorded for each trial. Each trial varies in terms of the amount of reward and the amount of time to wait. To model the decisions, a hyperbolic discounting function is generally used.
Inhibition and activation systems. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17)
  This will be assessed using the Punishment Sensitivity and Reward Sensitivity Questionnaire (PSRSQ) of 48 items. Responses in the scale are in a yes/no format. Higher punishment sensitivity scores are associated with lower number of punishable errors while higher reward sensitivity scores are linked to higher number of passive avoidance errors.
Self-reported impulsivity. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17)
  Impulsive behaviour scale (UPPS-P). Self-reported impulsivity will be measured with Impulsive behaviour scale (UPPS-P). It consists of 20 items scored on a four point Likert scale, ranging from strongly agree (1) to strongly disagree (4). Higher scores mean worse outcome in impulsivity, while lower scores are related to better self-control and regulation
Working Memory. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17)
  Working Memory: N-back Task will be assessed using N-back Task score based on accuracy and reaction times. Higher accuracy scores indicate stronger working memory and attention, while faster reaction times are linked to quicker processing speed and decision-making.
Cognitive flexibility. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17)
  The Wisconsin Card Sorting Test (WCST) requires sorting response cards with one of four stimulus cards, using feedback based on a rule. Wisconsin Card Sorting Test will be administered to measure shift strategy in response to changing contingencies. There are128 trials where more correct responses, fewer perseverative and non perseverative errors, and more completed categories (max 6) are related to better performance
Decision making. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17)
  Decision making: The Iowa Gambling Task (IGT) assess real-world decision-making in a lab settin using money rewards. Iowa Gambling Task will be used to assess decision-making using money rewards.

OTHER OUTCOMES:
Descriptive measures | Pre-treatment assessment (week 2)
  A socio-demographic questionnaire will be administered to examine age, education, gender, socio-economic variables and clinical variables to consider exclusion and inclusion criteria. All these variables are qualitative.
Depression Symptoms. Screening | Pre-treatment assessment (week 2)
  Beck Depression Inventory (BDI-II) The Beck Depression Inventory (BDI-II) will also be used to rule out major depressive symptoms as an exclusion criteria. The scores range from 0 to 63 points. Participants with a score higher than 29, indicative of severe symptoms, will be excluded.
Anxiety Symptoms. Screening | Pre-treatment assessment (week 2)
  Depression Anxiety and Stress Scale-21 (DASS-21) The anxiety subscale of the DASS-21 will also be used to rule out symptoms of major anxiety as an exclusion criterion. The scores for both subscales range from 0 to 21. Participants with a score higher than 8, indicative of severe symptoms, will be excluded from the study.
Eating and Weight Patterns. Screening | Pre-treatment assessment (week 2)
  Questionnaire on Eating and Weight Patterns-5 (QEWP-5): it is adapted to DSM-5 criteria and will be used to exclude people with binge eating problems and bulimia. The QEWP-5 is not scored on a traditional numerical scale like other psychological tests; instead, responses are used to identify the presence of eating disorder symptoms. Positive responses to key questions about the frequency of binge eating, compensatory behaviors, and emotional distress may indicate the presence of an eating disorder.
Using of Health Resources | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  The Health Resources Questionnaire asks how often and why people have needed medical care and medicines in the last 3 month to measure the impact of the intervention in terms of health uses. Fewer visits to health professionals will be indicative of improvement.
Motivation to change | Pre-treatment assessment (week 2)
  Motivation to change. The Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES 00) adapted to excess weight will be used to assess motivation to change habits. It has 18 items that score readiness to change in people with abusive food use with a five point Likert scale, ranging from strongly disagree (1) to strongly agree (5). Higher scores mean better outcome in relation to motivation to change, while higher scores on ambivalence suggest doubts about the motivation to change.
Previous treatment history | Pre-treatment assessment (week 2)
  History of previous treatment, from pharmacological or nutritional to psychological, should be recorded.
Quality of Life (Measures to calculate cost effectiveness, cost utility and budget impact analyses) | Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17)
  SF-36 Quality of Life Questionnaire: Using the tariff validated for Spain. The SF-36 (Short Form 36 Health Survey) is one of the most widely used questionnaires to measure health-related quality of life.
  It consists of 36 questions assessing eight key dimensions: physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role and mental health. Each dimension is scored on a scale of 0 to 100, where 0 represents the worst health status and 100 the best.
Years of Life Adjusted for Quality (Measures to calculate cost effectiveness, cost utility and budget impact analyses) | Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17)
  Years of Life Adjusted for Quality (QALY) is a measure used in healthcare to assess the value of medical treatments or interventions, combining quantity and quality of life. One QALY is equivalent to one year of life in full health. If a person lives a year with a reduced quality of life (due to illness, for example), a value of less than 1 is assigned, depending on the degree of well-being. This metric allows the effectiveness of different interventions to be compared, helping in health decision-making and resource allocation. It combines life years and quality (from SF-36) used in economic evaluation and cost-utility analyses of the intervention.
Binge Eating (BE) (Measures to calculate cost effectiveness, cost utility and budget impact analyses) | Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17)
  Changes in BE, assessed with BES for cost-effectiveness. The Binge Eating Scale (BES) (Escrivá-Martínez et al., 2019) is a self-administered questionnaire composed of 16 items: eight items that describe behavioral manifestations (for example, eating fast or consuming large amounts of food) and eight items on associated feelings and cognitions (for example, fear of not stopping eating). Each item has a response range from 0 to 3 points (0 = no severity of the symptom, 3 = serious problems on the symptom)
Intensity of Food Craving (Measures to calculate cost effectiveness, cost utility and budget impact analyses) | Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17)
  The FCQ-S-r will be used to assess the success of the intervention in the cost-effectiveness calculations.
Health Resource Costs (Measures to calculate cost effectiveness, cost utility and budget impact analyses) | Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17)
  Health Resource Costs: Includes visits to primary care, emergencies, hospital admissions, and medication costs. The Health Resource Questionnaire will be used to assess the success of the intervention in the cost-effectiveness calculations.
iTBS Session Staff Time (Measures to calculate cost effectiveness, cost utility and budget impact analyses) | Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17)
  Cost of a Clinical Psychology Area Specialist (FEA) for 3 minutes per session over 10 days, based on Andalusian Health Service remuneration will be used to assess the success of the intervention in the cost-effectiveness calculations.
Inhibitory Control Training Session Staff Time (Measures to calculate cost effectiveness, cost utility and budget impact analyses) | Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17)
  Training Session Staff Time: Cost of a Clinical Psychology Specialist (FEA) for 10 minutes per session over 10 days, based on Andalusian Health Service remuneration will be used to assess the success of the intervention in the cost-effectiveness calculations.
Equipment Costs (Measures to calculate cost effectiveness, cost utility and budget impact analyses) | Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17)
  Cost of fMRI and iTBS equipment will be used to assess the success of the intervention in the cost-effectiveness calculations.
Hormone levels (Biological samples collection) | Measured at Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17).
  Biological samples will be collected and deep-frozen in the CIMCYC until mass analyses are performed at the end of the project.
  Fasting blood tests will determine hormone levels (pg/ml) of estradiol, progesterone, cortisol, leptin, adiponectin, TSH, thyroxine, triiodothyronine, ghrelin, glucagon and GLP-1. A total of 10 ml of blood will be collected and centrifuged to separate the plasma from the rest and stored at -80ºC
Glucose and triglycerides levels (Biological samples collection) | Measured at Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17).
  Biological samples will be collected and deep-frozen in the CIMCYC until mass analyses are performed at the end of the project.
  Fasting blood tests will glucose and triglycerides levels (mg/dl). A total of 10 ml of blood will be collected and centrifuged to separate the plasma from the rest and stored at -80ºC
Insulin levels (Biological samples collection) | Measured at Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17).
  Biological samples will be collected and deep-frozen in the CIMCYC until mass analyses are performed at the end of the project.
  Fasting blood tests will determine insulin levels (U/ml). A total of 10 ml of blood will be collected and centrifuged to separate the plasma from the rest and stored at -80ºCa. Blood: Fasting blood tests will determine estradiol, progesterone, cortisol, leptin, adiponectin, TSH, thyroxine, triiodothyronine, ghrelin, glucagon, GLP-1, PYY (3-36), glucose, triglycerides, insulin, TNF-alpha, CRP, and IL-6. In addition, genetic analysis will be performed by sequencing candidate genes. A total of 10 ml of blood will be collected and centrifuged to separate the plasma from the rest and stored at -80ºC
Inflammatory parameters (Biological samples collection) | Measured at Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17).
  Biological samples will be collected and deep-frozen in the CIMCYC until mass analyses are performed at the end of the project.
  Fasting blood tests will determine IL-6, CRP, TNF-alpha levels (pg/ml). In addition, genetic analyseswill be performed by sequencing candidate genes. A total of 10 ml of blood will be collected and centrifuged to separate the plasma from the rest and stored at -80ºC
Satiety markers (Biological samples collection) | Measured at Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17).
  Biological samples will be collected and deep-frozen in the CIMCYC until mass analyses are performed at the end of the project.
  Fasting blood tests will determine PYY (3-36) levels (pg/ml). A total of 10 ml of blood will be collected and centrifuged to separate the plasma from the rest and stored at -80ºC
Genetic analyses (Biological samples collection) | Measured at Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17).
  Biological samples will be collected and deep-frozen in the CIMCYC until mass analyses are performed at the end of the project.
  Fasting blood tests will determine genetic analyses will be performed by sequencing candidate genes. Genome-wide association analysis is proposed to identify new genes and variants associated with PD such as ZFP36, GAD2 on chromosome 10p12, Neuromedin β with whole exome sequencing and methylation analysis.A total of 10 ml of blood will be collected and centrifuged to separate the plasma from the rest and stored at -80ºC
Oral microbiota (Biological samples collection) | Measured at Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17).
  Biological samples will be collected and deep-frozen in the CIMCYC until mass analyses are performed at the end of the project.
  Saliva samples for oral microbiota analyses will be collected using three swabs (right cheek, left cheek, tongue) that will be stored at -80ºC
Gut microbiota (Biological samples collection) | Measured at Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17).
  Biological samples will be collected and deep-frozen in the CIMCYC until mass analyses are performed at the end of the project.
  Participants will collect fecal samples and 1.5 g of the top layer will be stored in tubes at -80ºC for gut microbiota analyses.
Proteomics analysis. (Biological samples collection) | Measured at Pre-treatment assessment (week 2), post-treatment assessment (week 5) and follow-up (week 17).
  Biological samples will be collected and deep-frozen in the CIMCYC until mass analyses are performed at the end of the project.
  Samples for proteomics analyses will be collected in plastic bottles, centrifuged and stored at -80ºC

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Vilar-López, Ph.D, Principal Investigator — Universidad de Granada
Locations (1):
- Mind, Brain and Behavior Research Center at University of Granada (CIMCYC-UGR), Granada, Spain

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, will be shared.
Time Frame: Data will be available beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee and who provide a methodologically sound proposal. Proposals should be directed to rvilar@ugr.es

REFERENCES:
- [Background] Barone J, Oliveri M, Bonaventura RE, Mangano GR. Reduction of drive for thinness and body dissatisfaction in people with self-reported dysregulated eating behaviors after intermittent theta burst stimulation (iTBS) of the left dorsolateral prefrontal cortex. Front Hum Neurosci. 2023 Mar 17;17:1108869. doi: 10.3389/fnhum.2023.1108869. eCollection 2023. PMID 37007674
- [Background] Beam W, Borckardt JJ, Reeves ST, George MS. An efficient and accurate new method for locating the F3 position for prefrontal TMS applications. Brain Stimul. 2009 Jan;2(1):50-4. doi: 10.1016/j.brs.2008.09.006. PMID 20539835
- [Background] Chen T, Su H, Li R, Jiang H, Li X, Wu Q, Tan H, Zhang J, Zhong N, Du J, Gu H, Zhao M. A transcranial magnetic stimulation protocol for decreasing the craving of methamphetamine-dependent patients. STAR Protoc. 2021 Nov 10;2(4):100944. doi: 10.1016/j.xpro.2021.100944. eCollection 2021 Dec 17. PMID 34825214
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Kalla R, Muggleton NG, Cowey A, Walsh V. Human dorsolateral prefrontal cortex is involved in visual search for conjunctions but not features: a theta TMS study. Cortex. 2009 Oct;45(9):1085-90. doi: 10.1016/j.cortex.2009.01.005. Epub 2009 Feb 11. PMID 19269631
- [Background] Keeler JL, Chami R, Cardi V, Hodsoll J, Bonin E, MacDonald P, Treasure J, Lawrence N. App-based food-specific inhibitory control training as an adjunct to treatment as usual in binge-type eating disorders: A feasibility trial. Appetite. 2022 Jan 1;168:105788. doi: 10.1016/j.appet.2021.105788. Epub 2021 Oct 30. PMID 34728250
- [Background] Lawrence, N. S., Van Beurden, S., Javaid, M., & Mostazir, M. M. (2018). Mass dissemination of web and smartphone-delivered food response inhibition training to reduce unhealthy snacking. Appetite, 130, 309. https://doi.org/10.1016/j.appet.2018.05.207
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Escriva-Martinez T, Galiana L, Rodriguez-Arias M, Banos RM. The Binge Eating Scale: Structural Equation Competitive Models, Invariance Measurement Between Sexes, and Relationships With Food Addiction, Impulsivity, Binge Drinking, and Body Mass Index. Front Psychol. 2019 Mar 22;10:530. doi: 10.3389/fpsyg.2019.00530. eCollection 2019. PMID 30967808
- [Background] Meule A, Hermann T, Kubler A. A short version of the Food Cravings Questionnaire-Trait: the FCQ-T-reduced. Front Psychol. 2014 Mar 4;5:190. doi: 10.3389/fpsyg.2014.00190. eCollection 2014. PMID 24624116
- [Background] Neveu R, Neveu D, Carrier E, Gay A, Nicolas A, Coricelli G. Goal Directed and Self-Control Systems in Bulimia Nervosa: An fMRI Study. EBioMedicine. 2018 Aug;34:214-222. doi: 10.1016/j.ebiom.2018.07.012. Epub 2018 Jul 22. PMID 30045816
- [Background] Vioque J, Navarrete-Munoz EM, Gimenez-Monzo D, Garcia-de-la-Hera M, Granado F, Young IS, Ramon R, Ballester F, Murcia M, Rebagliato M, Iniguez C; INMA-Valencia Cohort Study. Reproducibility and validity of a food frequency questionnaire among pregnant women in a Mediterranean area. Nutr J. 2013 Feb 19;12:26. doi: 10.1186/1475-2891-12-26. PMID 23421854
- [Background] Daza, P., Novy, D. M., Stanley, M. A., & Averill, P. (2002). The Depression Anxiety Stress Scale-21: Spanish translation and validation with a Hispanic sample. Journal of Psychopathology and Behavioral Assessment, 24(3), 195-205. https://doi.org/10.1023/A:1016014818163
- [Background] Sanz, J., Navarro, M. E., y Vázquez, C. (2003). Adaptación española del Inventario para la Depresión de Beck-II (BDI-II): 1. Propiedades psicométricas en estudiantes universitarios. Análisis y Modificación de Conducta, 29, 239-288.
- [Background] Cebolla A, Barrada JR, van Strien T, Oliver E, Banos R. Validation of the Dutch Eating Behavior Questionnaire (DEBQ) in a sample of Spanish women. Appetite. 2014 Feb;73:58-64. doi: 10.1016/j.appet.2013.10.014. Epub 2013 Oct 28. PMID 24177441
- [Background] Mason AE, Vainik U, Acree M, Tomiyama AJ, Dagher A, Epel ES, Hecht FM. Improving Assessment of the Spectrum of Reward-Related Eating: The RED-13. Front Psychol. 2017 May 30;8:795. doi: 10.3389/fpsyg.2017.00795. eCollection 2017. PMID 28611698
- [Background] Burgess EE, Turan B, Lokken KL, Morse A, Boggiano MM. Profiling motives behind hedonic eating. Preliminary validation of the Palatable Eating Motives Scale. Appetite. 2014 Jan;72:66-72. doi: 10.1016/j.appet.2013.09.016. Epub 2013 Sep 25. PMID 24076018
- [Background] Gross, J. J., & John, O. P. (2003). Emotion Regulation questionnaire. En PsycTESTS Dataset. https://doi.org/10.1037/t06463-000
- [Background] Davidson EJ, Wright P. Selective processing of weight- and shape-related words in bulimia nervosa: use of a computerised Stroop test. Eat Behav. 2002 Autumn;3(3):261-73. doi: 10.1016/s1471-0153(02)00064-8. PMID 15001004
- [Background] Epstein LH, Salvy SJ, Carr KA, Dearing KK, Bickel WK. Food reinforcement, delay discounting and obesity. Physiol Behav. 2010 Jul 14;100(5):438-45. doi: 10.1016/j.physbeh.2010.04.029. Epub 2010 May 21. PMID 20435052
- [Background] Torrubia, R., Ávila, C., Moltó, J., & Caseras, X. (2001). The Sensitivity to Punishment and Sensitivity to Reward Questionnaire (SPSRQ) as a measure of Gray's anxiety and impulsivity dimensions. Personality And Individual Differences, 31(6), 837-862. https://doi.org/10.1016/s0191-8869(00)00183-5
- [Background] Lynam, D. R., Smith, G. T., Whiteside, S. P., & Cyders, M. A. (2006). The UPPS-P: Assessing five personality pathways to impulsive behavior. West Lafayette, IN: Purdue University, 10.
- [Background] KIRCHNER WK. Age differences in short-term retention of rapidly changing information. J Exp Psychol. 1958 Apr;55(4):352-8. doi: 10.1037/h0043688. No abstract available. PMID 13539317
- [Background] Grant, D. A., & Berg, E. A. (1948). Wisconsin card sorting Test. En PsycTESTS Dataset. https://doi.org/10.1037/t31298-000
- [Background] Bechara A, Damasio AR, Damasio H, Anderson SW. Insensitivity to future consequences following damage to human prefrontal cortex. Cognition. 1994 Apr-Jun;50(1-3):7-15. doi: 10.1016/0010-0277(94)90018-3. PMID 8039375
- [Background] Yanovski SZ, Marcus MD, Wadden TA, Walsh BT. The Questionnaire on Eating and Weight Patterns-5: an updated screening instrument for binge eating disorder. Int J Eat Disord. 2015 Apr;48(3):259-61. doi: 10.1002/eat.22372. Epub 2014 Dec 26. No abstract available. PMID 25545458
- [Background] Vieira da Silva R, de Oliveira IR, Lopes Velasquez M. Stages of Change Readiness and Treatment Eagerness Scale in Overweight and Obesity's Psychometric Properties (SOCRATES-OO). J Clin Psychol Med Settings. 2020 Dec;27(4):805-817. doi: 10.1007/s10880-019-09672-w. PMID 31667648
- [Background] Abellan Perpinan JM, Sanchez Martinez FI, Martinez Perez JE, Mendez I. Lowering the 'floor' of the SF-6D scoring algorithm using a lottery equivalent method. Health Econ. 2012 Nov;21(11):1271-85. doi: 10.1002/hec.1792. Epub 2011 Oct 4. PMID 21976290
- See also: Web of the project — http://trainep.ugr.es/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT06649994/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT06649994/ICF_001.pdf